CLINICAL TRIAL: NCT03535584
Title: Exercise as an Intervention to Treat Frailty and Decreased Physical Function in Kidney Transplant Candidates
Brief Title: Exercise to Treat Frailty and Decreased Physical Function in Transplant Candidates
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment was stopped due to covid-19 pandemic. An alternate study was initiated under an alternate IRB and clinical trial registration which allowed home exercise instead of in-center exercise after a prolonged pause in enrollment.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cassie C. Kennedy, M.D., Associate Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-009722
Record Dates: First submitted 2018-05-03; First posted 2018-05-24 (Actual); Last update posted 2025-03-31 (Actual); Status verified 2025-03

CONDITIONS: Kidney Transplant; Frailty
MeSH Terms: conditions — Frailty | interventions — Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Program (Experimental): All participants will attend a 16-session exercise program based on pulmonary rehabilitation and will complete questionnaires and frailty testing.
  Interventions: Behavioral: Exercise Program

INTERVENTIONS:
Behavioral: Exercise Program — Participants will be asked to complete 2 1-hour exercise sessions per week for 8 weeks (16 total sessions) under the supervision of a licensed respiratory therapist on non-dialysis days. The exercise program will be based on pulmonary rehabilitation and will follow guidelines established by the American Thoracic Society. Exercise sessions will include endurance (treadmill or cycle ergometer), strength (weight resistance), and flexibility training. Exercise sessions will be tailored to individual participants, and participant safety will be monitored during each session.

SUMMARY:
Frailty is a condition characterized by slowness, weakness, low physical activity, wasting, and exhaustion. Frailty increases the risk for adverse outcomes following transplant such as increased length of stay in the hospital, mortality, or graft function. No interventions for frailty are known for patients with renal disease, but exercise programs like pulmonary rehabilitation have been effective in improving frailty in patients with other diseases, such as lung disease. The goal of this study is to test whether exercise will also improve frailty among patients who are waiting for a kidney transplant and who are considered frail or pre-frail.

DETAILED DESCRIPTION:
RECRUITMENT: This study will be conducted at Mayo Clinic in Rochester, MN. Patients over 18 who have chronic kidney disease will be approached for recruitment. Interested patients will go through the informed consent process and, if frailty testing was not completed within the two weeks prior to consent, patients will complete frailty testing. If patients are considered frail or pre-frail, they will be enrolled in the study.

FRAILTY TESTING: Participants will complete the FP, Short Physical Performance Battery (SPPB) and other frailty testing at the beginning of the study, 4 weeks after beginning the intervention, and 8 weeks after beginning the intervention. Frailty testing will include a hand grip strength test, a gait speed test over 15 feet, repeated chair stands, balance testing, and a body composition scan. Participants will also be asked to wear an activity monitor for 5-7 days at each testing point and to complete a set of questionnaires. Height, weight, BMI, skeletal muscle mass, percent body fat, and segmental lean mass will be recorded. Participants with a pacemaker, an implantable cardioverter-defibrillator (ICD), or an automated ICD (AICD) will not be able to complete. At enrollment, participants 55 and older will undergo a submaximal exercise test to rule out significant undiagnosed cardiopulmonary disease (standard entrance criteria for pulmonary rehabilitation).

INTERVENTION: Participants will be asked to complete 2 1-hour exercise sessions per week for 8 weeks (16 total sessions) under the supervision of a licensed respiratory therapist in Rochester, MN on non-dialysis days unless the participant is on daily or near-daily dialysis (e.g. home hemodialysis or peritoneal dialysis). . The exercise sessions will be based on pulmonary rehabilitation and will follow guidelines established by the American Thoracic Society. Exercise sessions will include endurance (treadmill or cycle ergometer), strength, and flexibility training and will be tailored to individual participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Consenting to research
* CKD (stages 1-5)
* An SPPB score ≤10 or considered frail or pre-frail by FP

Exclusion Criteria:

* Younger than 18 years
* Patients listed for heart or lung transplants
* Terminal illness with a prognosis of less than 6 months
* Significant comorbidities that limit rehabilitation potential including pulmonary disease requiring continuous oxygen supplementation, active angina, critical aortic sclerosis, decompensated heart failure, or known ventricular arrhythmia.
* Kidney transplant candidates without cardiac clearance for transplant
* An SPPB score >10 or not considered frail or pre-frail by FP
* Non-English speaker without availability of adequate interpreter services (safety concern)
* Failure to pass submaximal exercise test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Change in Frailty Status | 2 Months
  Frailty will be determined by Frailty Phenotype (FP) or Short Physical Performance Battery (SPPB) scores. FP is determined by the presence of 3 or more of the following: slowness (measured by gait speed), exhaustion (measured with the CES-D), weakness (measured by hand grip strength), low physical activity level (measured with the MLTPAQ and activity monitoring), and wasting (measured through self-report or by tracking changes in weight). The SPPB consists of a gait speed test, balance testing, and repeated chair stands. A score less than or equal to 10 will be considered frail.

SECONDARY OUTCOMES:
Change in Grip Strength | 2 Months
  Hand grip strength will be measured using a hand-held dynamometer. Frailty is characterized as the lowest 20% by gender and body mass index.
Change in Gait Speed | 2 Months
  Gait speed will be measured over a distance of 15 feet at the patient's self-selected walking speed. Frailty is characterized as the slowest 20% by gender and height. Results will be prorated for 4 meters for the SPPB score.
Change in Exhaustion | 2 Months
  Patients will self-report their level of exhaustion using the Center for Epidemiologic Studies Depression Scale (CES-D) which consists of a 4-point scale. Items on the CES-D are scored from minimum to maximum values (1 point to 4 points) which are indicated on the CES-D as "rarely or none of the time," "some or a little of the time," "occasionally or a moderate amount of time," "most or all of the time," respectively. A higher number of points indicates a worse outcome.
Change in Activity | 2 Months
  Energy expenditure will be measured using an activity monitor worn on the wrist for 5-7 days. Low activity is defined as activity in the lowest 20% (<383 Kcals/week for men or <270 Kcals/week for women). Patients will also self-report their activity level using the MLTPAQ.
Wasting | 2 Months
  Wasting is defined as a decrease in lean body mass or unintentional weight loss of 10 or more pounds in one year.
Change in SPPB Score | 2 Months
  The SPPB consists of a gait speed test, repeated chair stands, and balance testing. Lower scores indicate decreased physical function.
Change in Quality of Life | 2 Months
  Health-related quality of life will be measured using the KDQOL-SF.
Post-Transplant Outcomes | 1 Year
  The relationship between exercise, frailty status, and post-transplant outcomes will be examined for patients who receive a transplant within 1 year of enrolling in this study. The various outcome measures will be aggregated to indicate mortality rate up to one year post-transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Cassie C Kennedy, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lorenz EC, Hickson LJ, Hogan MC, Kennedy CC. Examining the safety and effectiveness of a 4-week supervised exercise intervention in the treatment of frailty in patients with chronic kidney disease. Clin Kidney J. 2023 Aug 9;16(11):2003-2010. doi: 10.1093/ckj/sfad192. eCollection 2023 Nov. PMID 37915911
- [Derived] Lorenz EC, Hickson LJ, Weatherly RM, Thompson KL, Walker HA, Rasmussen JM, Stewart TL, Garrett JK, Amer H, Kennedy CC. Protocolized exercise improves frailty parameters and lower extremity impairment: A promising prehabilitation strategy for kidney transplant candidates. Clin Transplant. 2020 Sep;34(9):e14017. doi: 10.1111/ctr.14017. Epub 2020 Jul 24. PMID 32573816